CLINICAL TRIAL: NCT01303432
Title: Double-blind, Placebo-controlled Nutrition Intervention Trial, to Study Efficacy and Safety of Yogurts Supplemented With Mobilee on Joint Function, Joint Structure and Quality of Life of Adults With Low Intensity Gonalgia
Brief Title: Effect of Yogurts Supplemented With Mobilee on Joint Function in Healthy Individuals With Joint Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioiberica (Industry)
Collaborators: Technological Centre of Nutrition and Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CTNS 001_03_2010
Record Dates: First submitted 2011-02-21; First posted 2011-02-24 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Low Intensity Knee Gonalgia
Keywords: Joint discomfort; Functional Food; Joint function; Mobilee
MeSH Terms: interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobilee yogurt (Experimental): Subjects eating daily on yogurt supplemented with Mobilee
  Interventions: Dietary Supplement: Yogurt supplemented with Mobilee
- Placebo yogurt (Placebo Comparator): Subjects receiving daily a standard yogurt
  Interventions: Dietary Supplement: Yogurt

INTERVENTIONS:
Dietary Supplement: Yogurt supplemented with Mobilee — One yogurt (125mL) per day including 80mg of Mobilee
  Arms: Mobilee yogurt
Dietary Supplement: Yogurt — One yogurt (125mL) per day
  Arms: Placebo yogurt

SUMMARY:
The purpose of this study is to determine whether the daily eating of a yogurt supplemented with Mobile is effective in improving joint function and quality of life of individuals with low intensity gonalgia.

DETAILED DESCRIPTION:
The prevalence of low intensity gonalgia is relatively high in western population. The purpose of the present intervention study is to determine whether the daily consumption of a yogurt supplemented with Mobile is effective in improving joint function and quality of life of individuals with low intensity gonalgia. Previous research using in vitro and animal models have demonstrated the efficacy of Mobilee in reducing inflammation and promoting anabolic responses in joint tissues. In addition, in two previous human intervention trials, the effects of Mobilee in joint function had been assessed using isokinetic tests. The present trial aims to confirm those previous results.

ELIGIBILITY:
Inclusion Criteria:

* Adult (between 20 and 70 years of age)
* Subject with low intensity knee gonalgia (VAS pain intensity between 3 and 5cm during at least the last 6 months)
* Healthy individual according to its medical records, physical and laboratorial parameters
* Positive informed consent

Exclusion Criteria:

* Individuals requiring acetaminophen or any other drug to control pain
* Active rheumatoid arthritis or any other inflammatory joint disease
* Oral treatment with corticosteroids 4 weeks before selection
* Intra-articular treatment with corticosteroids 3 months before selection
* Significant injury of the study joint 12 months before selection
* Individuals receiving any drug or supplement for osteoarthritis
* Individuals requiring any type of medical prescription to control pain

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in isokineic assessment of muscular strength | 3 months
  The muscular isokinetic assessment determines peak torque, power mean and total work of a certain joint using a dynamometric computerized system. The principal parameter is the change from baseline in the peak torque of the affected joint in extension at a speed of 240º/sec measured in Nm (Newton-meter).

SECONDARY OUTCOMES:
Change from baseline in isokinetic assessment of muscular strength (other conditions) | 3 months
  Change from baseline of peak torque (Nm), power mean (W) and total work (J) of the affected joint in extension at 180º/sec, and in flexion at 240º/sec and 180º/sec.
Assessment of joint swelling, effusion | 3 months
  Ultrasonography: Study of the synovial effusion degree (if any) measured in the longitudinal axis of the suprapatellar recess of the affected knee.Results are expressed as change from baseline in mm.
Pain assessment (VAS) | 3 months
  Time evolution of pain intensity as measured by Visual Analogue Scale (mm).
SF-36 Health questionnaire | 3 months
  Questionnaire SF36-v2 to measure physical and mental health.
Number of Participants with Adverse Events | 3 months
  The safety assessment includes a register of the appearance of adverse events along the 3 months of the study
Subjective evaluation of the intervention | 3 months
  Questionnaire to evaluate the subjective perception of the efficacy of the intervention.
Change from baseline in systolic blood pressure, hearth rate, general biochemical profile and body mass index at 3 months | 3 months
  Safety assessment includes an evaluation at 3 months of changes from baseline on systolic blood pressure, hearth rate, general biochemical profile and body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, MD, Principal Investigator — Hospital Universitari Sant Joan de Reus
Locations (1):
- Hospital Universitari Sant Joan de Reus, Reus, Tarragona, Spain

REFERENCES:
- See also: Related Info — http://www.cdti.es/